CLINICAL TRIAL: NCT06094725
Title: An Open-label, Multiple-dose, Adaptive Design Study to Evaluate the Effects of Hepatic Impairment on the Pharmacokinetics of Relacorilant
Brief Title: A Study to Evaluate the Effects of Hepatic Impairment on the Pharmacokinetics of Relacorilant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CORT125134-128
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- No Hepatic Impairment (Experimental): Subjects with no hepatic impairment will receive relacorilant 300 mg once daily on Days 1 through 10.
  Interventions: Drug: Relacorilant
- Moderate Hepatic Impairment (Experimental): Subjects with moderate hepatic impairment (Child-Pugh Class B) will receive relacorilant 300 mg once daily on Days 1 through 10.
  Interventions: Drug: Relacorilant
- Mild Hepatic Impairment (Experimental): Subjects with mild hepatic impairment (Child-Pugh Class A) will receive relacorilant 300 mg once daily on Days 1 through 10.
  Interventions: Drug: Relacorilant

INTERVENTIONS:
Drug: Relacorilant — Relacorilant 300 mg (3 X 100 mg softgel capsules) for oral administration
  Other Names: CORT125134

SUMMARY:
The primary objective of this multiple-dose, adaptive design study is to evaluate the effect of hepatic impairment on the pharmacokinetics (PK) of relacorilant relative to healthy matched control male and female subjects (Part 1).

DETAILED DESCRIPTION:
If an obvious effect of moderate hepatic impairment on exposure to relacorilant is observed in Part 1, optional Part 2 of the study will be conducted. In Part 2, the effect of mild hepatic impairment on the PK of relacorilant will be evaluated, using control data from the same healthy control subjects who were matched to the subjects in Part 1.

Secondary objectives of the study are 1) evaluation of the effect of hepatic impairment on the PK of relacorilant metabolites, and 2) evaluation of safety and tolerability of relacorilant on healthy subjects and those with hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the purpose and risks of the study and is willing and able to adhere to scheduled visits, treatment plans, laboratory tests, and other study evaluations and procedures
* Provide written informed consent before any study-specific procedure is performed
* Male or a nonpregnant, nonlactating female judged to be in good health, except for allowance of health conditions consistent with hepatic impairment
* Body mass index (BMI) between 18 and 32 kg/m^2, inclusive, and a body weight more than 50 kg (110 pounds)
* Estimated glomerular filtration rate (eGFR) ≥80 mL/minute/1.73 m^2
* Suitable veins for multiple venipuncture/cannulation
* Agrees to limit smoking or use of tobacco or nicotine-containing products to less than 5 cigarettes or uses per day
* Willing to comply with study restrictions as described in the protocol
* Female subject is of either nonchildbearing potential (ie, postmenopausal or permanently sterilized) or uses highly effective contraception with low user-dependency, as described in the protocol.

Subjects with normal hepatic function must also satisfy the following inclusion criteria:

* Clinical laboratory results within the reference range at Screening and Day -1, unless considered not clinically significant by the Principal Investigator
* Negative screening results for hepatitis B surface antigen, hepatitis C virus antibody, and HIV antibodies.

Subjects with moderate or mild hepatic impairment must also satisfy the following inclusion criteria:

* Documented parenchymal hepatic disease
* Liver dysfunction of moderate (Child-Pugh Class B [score of 7 to 9]; Part 1) or mild (Child-Pugh Class A [score of 5 to 6]; Part 2) severity
* Stable hepatic impairment defined as no clinically significant change in disease status within the last 30 days
* On a stable dose of medication and/or treatment regimen at least 2 weeks before study drug dosing
* If a subject has nonhepatic abnormal clinical laboratory results, these results are considered not clinically relevant by the Principal Investigator (or designee) and the medical monitor.

Exclusion Criteria:

* An employee or immediate family member of the Clinical Research Unit (CRU) or the Sponsor
* Has been previously enrolled in any study of relacorilant
* Has multiple clinically significant drug allergies or is allergic to any of the components of relacorilant
* Has a condition that could be aggravated by excessive glucocorticoid receptor antagonism. Subjects with inactive seasonal hay fever or childhood asthma may be included.
* Has a history of malabsorption syndrome or previous gastrointestinal surgery that could affect drug absorption or metabolism
* Has Gilberts syndrome
* Has current or previous (within a 1-year period) alcohol or substance abuse and/or dependence
* Has evidence of acute viral hepatitis in the 3 calendar months before the first dose of study drug
* In the 2 calendar months before the first dose of study drug, subject has: donated/lost blood or plasma in excess of 400 mL, or received an investigational drug
* Has a positive result for alcohol or drugs of abuse at Screening or upon admission to the CRU
* Has clinically relevant abnormal vital signs, physical examination, laboratory tests, or 12-lead ECG findings at Screening and/or before the first dose of study drug, other than those associated with chronic hepatic impairment
* Has taken any prohibited prior medication, as described in the protocol
* Has any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Principal Investigator.

Additional exclusion criteria for subjects with moderate or mild hepatic impairment:

* Has hepatic encephalopathy of Grade 2 that has not been controlled with medication for the previous 3 calendar months before Screening or of Grade 3 or higher within the previous 3 calendar months before Screening, regardless of use of medication for the treatment of hepatic encephalopathy
* Has a history of liver transplantation, hepatocellular carcinoma, portosystemic shunt, or acute liver disease (eg, caused by infection or drug toxicity).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of plasma relacorilant during the dosing interval (Cmax) | Predose and at serial time points up to 24 hours after dosing on Day 10
Area under the concentration-time curve of plasma relacorilant from time zero to the end of the dosing interval (24 hours) (AUCt) | Predose and at serial time points up to 24 hours after dosing on Day 10

SECONDARY OUTCOMES:
Cmax of relacorilant plasma metabolites | Predose and at serial time points up to 24 hours after dosing on Day 10
AUCt of relacorilant plasma metabolites | Predose and at serial time points up to 24 hours after dosing on Day 10
Number of subjects with one or more treatment-emergent adverse events | Up to Day 20
Number of subjects with one or more treatment-emergent adverse events by severity | Up to Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Custodio, Study Director — Corcept Therapeutics
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No